CLINICAL TRIAL: NCT06711978
Title: Comparison of the Efficacy and Safety of Mirogabalin and Duloxetine in Chemotherapy-induced Peripheral Neuropathy in a Randomized Controlled Trial: a Quality of Life Study in Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-2024-072
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: CIPN; CIPN - Chemotherapy-Induced Peripheral Neuropathy; CIPN in Adjuvant Breast Cancer Patients; Duloxetine; Mirogabalin
MeSH Terms: interventions — mirogabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirogabalin Group (Experimental)
  Interventions: Drug: Duloxetine
- Duloxetine Group (Active Comparator)
  Interventions: Drug: Mirogabalin

INTERVENTIONS:
Drug: Mirogabalin — Participants will receive Mirogabalin at a dose of twice daily for 4 weeks to manage CIPN pain.
  Arms: Duloxetine Group
Drug: Duloxetine — Participants will receive Duloxetine at a dose of once daily for 4 weeks to manage CIPN pain.
  Arms: Mirogabalin Group

SUMMARY:
To conduct a two-arm, parallel, prospective, randomized controlled, open-label trial to compare the efficacy of the novel drug mirogabalin with the conventional treatment duloxetine in reducing pain associated with chemotherapy-induced peripheral neuropathy (CIPN).

There will be a difference in pain reduction after 4 weeks of treatment between the mirogabalin group and the duloxetine group in patients with chemotherapy-induced peripheral neuropathy (CIPN).

Participants will:

* Take drug duloxetine or a mirogabalin every day for 4 weeks.
* Visit the clinic once every 2 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors aged 19 years or older.
* Peripheral, symmetrical pain in both feet occurring within 12 weeks of initiating chemotherapy with taxane or platinum agents (or their combination).
* Patients experiencing at least grade 2 peripheral neuropathy as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with an average pain intensity of 4 or higher on the Numerical Rating Scale (NRS) during the past week, following the completion of chemotherapy.
* Concurrent use of selected analgesics (acetaminophen, nonsteroidal anti-inflammatory drugs [NSAIDs]) is permitted if the following conditions are met:

  1. No new analgesics are introduced.
  2. Current analgesics are not discontinued.
  3. The total weekly 24-hour dose of analgesics does not vary by more than 10% during the 2 weeks prior to enrollment.
* Ongoing treatment for peripheral neuropathy or neuropathic pain must be discontinued at least 7 days before randomization

Exclusion Criteria:

* Patients with a prior diagnosis of peripheral neuropathy due to diabetes, trauma, alcohol abuse, compression, or other causes, or those with a previously diagnosed central nervous system disorder. (Patients with pre-existing diabetes or thyroid disease who had no symptoms of peripheral neuropathy, such as numbness or tingling in the hands or feet, before chemotherapy may be included.)
* Patients with significant psychiatric disorders, such as severe depression, bipolar disorder, or suicidal ideation.
* Pregnant or breastfeeding patients.
* Patients with a history of prior treatment with other neurotoxic chemotherapeutic agents.
* Patients with renal impairment (creatinine clearance < 30 mL/min) or hepatic dysfunction.
* Patients with planned surgical procedures within 4 weeks of enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form (BPI-SF) | From enrollment to the end of treatment at 4 weeks

SECONDARY OUTCOMES:
NCI-CTCAE v5.0 | From enrollment to the end of treatment at 4 weeks.
EORTC-QLQ-CIPN20 | From enrollment to the end of treatment at 4 weeks.
EORTC QLQ-C30 | From enrollment to the end of treatment at 4 weeks.
Korean neuropathic pain questionnaire neuropathic pain questionnaire(KPNQ) | From enrollment to the end of treatment at 4 weeks.
sural SNAP amplitude | At Baseline
peroneal cMAP amplitude | At Baseline
Medication compliance & ADRs | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yangsan Pusan National University Hospital, Mulgeum, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sundar R, Bandla A, Tan SS, Liao LD, Kumarakulasinghe NB, Jeyasekharan AD, Ow SG, Ho J, Tan DS, Lim JS, Vijayan J, Therimadasamy AK, Hairom Z, Ang E, Ang S, Thakor NV, Lee SC, Wilder-Smith EP. Limb Hypothermia for Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Study. Front Oncol. 2017 Jan 10;6:274. doi: 10.3389/fonc.2016.00274. eCollection 2016. PMID 28119855
- [Result] Misawa S, Denda T, Kodama S, Suzuki T, Naito Y, Kogawa T, Takada M, Suichi T, Shiosakai K, Kuwabara S; MiroCIP study group. Efficacy and safety of mirogabalin for chemotherapy-induced peripheral neuropathy: a prospective single-arm trial (MiroCIP study). BMC Cancer. 2023 Nov 11;23(1):1098. doi: 10.1186/s12885-023-11560-4. PMID 37951905
- [Result] Jordan B, Jahn F, Sauer S, Jordan K. Prevention and Management of Chemotherapy-Induced Polyneuropathy. Breast Care (Basel). 2019 Apr;14(2):79-84. doi: 10.1159/000499599. Epub 2019 Apr 10. PMID 31798378
- [Result] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Result] Hertz DL, Childs DS, Park SB, Faithfull S, Ke Y, Ali NT, McGlown SM, Chan A, Grech LB, Loprinzi CL, Ruddy KJ, Lustberg M. Patient-centric decision framework for treatment alterations in patients with Chemotherapy-induced Peripheral Neuropathy (CIPN). Cancer Treat Rev. 2021 Sep;99:102241. doi: 10.1016/j.ctrv.2021.102241. Epub 2021 Jun 9. PMID 34174668
- [Result] Loprinzi CL, Lacchetti C, Bleeker J, Cavaletti G, Chauhan C, Hertz DL, Kelley MR, Lavino A, Lustberg MB, Paice JA, Schneider BP, Lavoie Smith EM, Smith ML, Smith TJ, Wagner-Johnston N, Hershman DL. Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy in Survivors of Adult Cancers: ASCO Guideline Update. J Clin Oncol. 2020 Oct 1;38(28):3325-3348. doi: 10.1200/JCO.20.01399. Epub 2020 Jul 14. PMID 32663120